CLINICAL TRIAL: NCT05954286
Title: Master Protocol for Early Treatment and Post-Exposure Prophylaxis of COVID-19 Adaptive Platform Trial PROTECT-APT 1
Brief Title: PROTECT-APT 1: Early Treatment and Post-Exposure Prophylaxis of COVID-19
Acronym: PROTECT-APT 1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Henry M. Jackson Foundation for the Advancement of Military Medicine (Other)
Collaborators: Joint Program Executive Office Chemical, Biological, Radiological, and Nuclear Defense Enabling Biotechnologies (Other Government); RedHill Biopharma Limited (Industry); FHI Clinical, Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: PC06
Record Dates: First submitted 2022-03-30; First posted 2023-07-20 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-04

CONDITIONS: SARS-CoV-2
Keywords: COVID-19; Early Treatment; Post-Exposure Prophylaxis; Outpatient
MeSH Terms: conditions — COVID-19 | interventions — upamostat

STUDY DESIGN:
Intervention Model Description: An adaptive, randomized, double-blind, platform trial
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Early Treatment: Upamostat 400 mg (Experimental): 400 mg (2 x 200 mg) capsules administered orally once daily for 14 days
  Interventions: Drug: Upamostat
- Early Treatment: Placebo Oral Capsule (Placebo Comparator): The placebo arm may be pooled across more than one experimental arm if multiple investigational drug are available to be tested at the same time and administered in the same way.
  Interventions: Drug: Placebo (PO)

INTERVENTIONS:
Drug: Upamostat — Upamostat is available as a hydrogen sulphate salt (also designated as WX-671.1). WX-671.1 is a white to yellowish powder which is freely soluble in dimethyl sulfoxide and soluble in ethanol. The drug substance is very slightly soluble in water or 0.1 M HCl.
  Other Names: WX-671; RHB-107
  Arms: Early Treatment: Upamostat 400 mg
Drug: Placebo (PO) — Oral Capsules
  Arms: Early Treatment: Placebo Oral Capsule

SUMMARY:
This study is an adaptive, randomized, double blind, platform trial evaluating promising investigational products (IP) for safety and efficacy as early outpatient treatment and post-exposure prophylaxis for Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2).

DETAILED DESCRIPTION:
This multicenter trial will be conducted in both domestic and international sites. The study will compare IPs to control in standard and intermediate risk, non-hospitalized adult SARS-CoV-2 infected participants and uninfected adult contacts of SARS-CoV-2 confirmed cases. The master protocol will outline the core elements of the study. Investigational products may be included in either or both study indications: early treatment and post-exposure prophylaxis (PEP). The study includes a phase 2 evaluation for all IPs. The platform trial design will allow for multiple IPs to be incorporated into the protocol as product specific appendices (PSA) as products are identified and become available. Each PSA will detail the interventions, the endpoints, target treatment effect, intended statistical analysis, the relevant control arms, and the sample size range. The PSA may define additional adaptive design elements, such as early declaration rules.

ELIGIBILITY:
Population A: Symptomatic adults seeking care or testing for COVID-19

Inclusion Criteria:

1. Age ≥ 18 years
2. Positive molecular or antigen diagnostic test for SARS-CoV-2 at study enrollment or within ≤ 5 days prior to enrollment
3. Presence of two or more Screening Symptoms listed in Supplement 3 with at least two symptoms classified as moderate to severe (and/or ≥ 2 on the frequency questions or loss of taste/smell questions) at the time of enrollment a. For participants who have preexisting conditions causing mild or moderate symptoms listed on the Screening Symptom Questionnaire, there must be an increase of at least one severity level for that symptom at enrollment (For example, prior to illness participant routinely experienced headaches rated as moderate severity, now rating headache as severe at enrollment)

   * Supplement 3 Screening Symptoms: stuffy or runny nose, hoarse voice, sore throat, difficulty breathing, cough, fatigue (low energy or tiredness), muscle or body aches, headache, fever (documented temperature > 38° C [100.4° F]) or subjective fever, chills or shivering, feeling hot or feverish, nausea, vomiting, diarrhea, loss of smell, loss of taste
4. Symptom onset ≤ 5 days prior to enrollment

Exclusion Criteria:

1. Hospital admission at the time of enrollment
2. Hospitalization will be defined as requiring medical care not available in an outpatient setting for greater than 24 hours
3. Hospitalization for isolation or quarantine requirements or for social reasons will NOT constitute an exclusion criterion
4. Laboratory confirmed SARS-CoV-2 infection 6 to 90 days prior to enrollment
5. Oxygen saturation < 92% on room air
6. Baseline use of supplemental oxygen at the time of enrollment
7. Presence of any of the following comorbidities that per the PI puts the patient at high risk of developing severe COVID-19 illness:

   a. Age ≥ 75 years b. Active treatment for solid tumor and hematologic malignancies c. Hematologic malignancy, myeloma, or related disorder (e.g., myelodysplastic syndrome, myelofibrosis) d. Receipt of solid-organ transplant or an islet transplant and taking immunosuppressive therapy e. Chemotherapy or radiotherapy for solid organ cancer in the last 12 months f. Receipt of chimeric antigen receptor (CAR)-T-cell therapy or hematopoietic stem cell transplant (within 2 years of transplantation or taking immunosuppressive therapy) g. Moderate or severe primary immunodeficiency (e.g., common variable immunodeficiency disease, severe combined immunodeficiency, DiGeorge syndrome, Wiskott-Aldrich syndrome) h. Advanced or untreated HIV infection (people with HIV and CD4 cell counts less than 200/mm3, history of an AIDS-defining illness without immune reconstitution, or clinical manifestations of symptomatic HIV) i. Active treatment with high-dose corticosteroids (i.e., 20 or more mg of prednisone or equivalent per day when administered for 2 or more weeks), alkylating agents, antimetabolites, transplant-related immunosuppressive drugs, cancer chemotherapeutic agents classified as severely immunosuppressive, tumor necrosis factor (TNF) blockers, and other biologic agents that are immunosuppressive or immunomodulatory j. Sickle cell disease k. Chronic liver disease (e.g., Child-Pugh Class A, B or C cirrhosis) l. Down syndrome m. Dementia or neurocognitive disability (e.g., Parkinson's disease) n. Participants with 3 or more of the following conditions: i) No prior COVID-19 infection OR has not completed a COVID-19 vaccine series within the last 6 months OR has not received a vaccine booster within the last 6 months ii) Age 65-74 years iii) BMI ≥35 (or >95th percentile in adolescents) iv) Type 1 or type 2 diabetes mellitus v) Cardiovascular disease (including HTN if age >55) vi) Chronic lung disease (including bronchiectasis, CF, COPD, ILD, PHTN, PE, moderate-to-severe asthma) vii) Chronic kidney disease (eGFR <30)
8. Participants who are receiving or plan to receive anti-SARS-CoV-2 antivirals for treatment of their COVID-19

Population B: Uninfected adult contacts of symptomatic SARS-CoV-2 infected individuals

Inclusion Criteria:

1. Age ≥ 18 years
2. Asymptomatic contact of an individual with laboratory confirmed SARS-CoV-2 infection defined as:

   a. Indoor exposure to the symptomatic case or cases within 6 feet (2 meters) for ≥ 15 minutes over a 24-hour period without the use of personal protective equipment
3. Negative screening SARS-CoV-2 molecular or antigen diagnostic test performed at screening or within less than or equal to 24 hours of enrollment
4. Exposure and enrollment within 6 days or less from when the symptomatic, confirmed SARS-CoV-2 positive case first had symptoms

Exclusion Criteria:

1. Symptoms attributed to COVID-19 as assessed by the investigator 2. Positive molecular or antigen diagnostic test for SARS-CoV-2 from any upper respiratory specimen within 90 days prior to enrollment 3. SARS-CoV-2 vaccination within 90 days prior to enrollment EXCEPT if severely immunocompromised or a known vaccine non-responder 4. Severely immunocompromised or a known vaccine non-responder defined as: solid organ or stem cell transplant recipient, B cell leukemia, receiving B cell depletion therapy (e.g., rituximab), agammaglobulinemia, or negative serology ≥2 weeks after vaccination with two doses of a vaccine 5. Hospital admission at the time of enrollment

1. Hospitalization will be defined as requiring medical care not available in an outpatient setting for greater than 24 hours 6. Hospitalization for isolation or quarantine requirements or for social reasons will NOT constitute an exclusion criterion

   For Both populations:

   Inclusion Criteria:

   1. Must also meet the intervention specific inclusion/exclusion criteria for at least one PSA that is enrolling participants

   Exclusion Criteria:
   1. Absence of informed consent
   2. Pregnancy
   3. Breastfeeding
   4. Individuals who the study investigators believe are unable to comply with the requirements of the study
   5. Participation in another intervention trial for the treatment or prophylaxis of SARS-CoV-2 infection or COVID-19 disease at the time of enrollment

   Additional Criteria for the Early Treatment Upamostat Arm:

   Inclusion Criteria:

   1. Women of childbearing potential must agree to use an effective contraceptive method upon enrollment in the study through 8 weeks after the last dose of the investigational product. This would include oral contraceptives, implanted contraceptives, intrauterine devices, and barrier methods.

   - A woman is considered of childbearing potential unless post-menopausal (subject is at least 50 years old and has a history of ≥ 2 years without menses without other known or suspected cause), or permanently surgically sterilized.
   * Participants not of reproductive potential are eligible without requiring the use of a contraceptive method. Participant-reported history is acceptable documentation of surgical sterilization and menopause.

   Exclusion Criteria:

   1. Patient is currently taking or is expected to start taking warfarin, apixaban (Eliquis), or rivaroxaban (Xarelto). Patients may be taking or start on study dabigatran (Pradaxa), standard or low molecular weight heparin.

   2. Patients with prolonged QT/QTc interval and/or increased susceptibility to arrythmia defined as the presence of any of the following:

   - QTc interval > 450 msec

   - Pathological Q-waves (defined as Q-wave > 40 msec or depth > 0.4-0.5 mV)

   - Evidence of ventricular pre-excitation

   - Electrocardiographic evidence of complete LBBB, RBBB, incomplete LBBB, in complete RBBB

   - Evidence of second- or third-degree heart block
   * Intraventricular conduction delay with QRS duration > 120 msec
   * Bradycardia as defined by sinus rate< 50 bpm
   * Personal or family history of long QT syndrome
   * Personal history of cardiac disease, symptomatic or asymptomatic arrhythmias, except for sinus arrhythmia
   * Syncopal episodes or additional risk factors for torsades de points (e.g., heart failure, hypokalemia)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2024-01-29 (Actual); Primary Completion 2025-04-24 (Actual); Study Completion 2025-04-24 (Actual)

PRIMARY OUTCOMES:
Early Treatment: Time to sustained alleviation or resolution of COVID-19 symptoms | Day 0 to Day 28
  Defined as the number of days from randomization within a PSA to the first day the participant reports all symptoms as mild or none for at least 3 consecutive days. Symptoms will be assessed via completion of a Screening Symptom Questionnaire at Enrollment and then a Daily Follow Up Symptom Questionnaire.
Post-Exposure Prophylaxis: Incidence of symptomatic COVID-19 by Day 14 | Day 0 to Day 14
  Defined as a positive SARS-CoV-2 RT-PCR test and the presence of at least one COVID-19 symptom. COVID-19 symptoms will be ascertained using the Daily Follow Up Symptom Questionnaire.

SECONDARY OUTCOMES:
Early Treatment: Number and proportion of all cause hospitalizations | Day 0 to Week 12
Early Treatment: Number and proportion of all cause deaths | Day 0 to Week 12
Early Treatment Upamostat Arm: Change in overall COVID-19 symptom severity score | Day 0 to Day 28
  A mixed model repeated measure (MMRM) model will be used to model the symptom severity score at each day using the baseline symptom score, participant, day, and treatment by day as covariates.
Early Treatment Upamostat Arm: Proportion of participants in each treatment group developing new COVID-19 symptoms rated as severe | Day 0 to Day 28
  A Cox proportional hazards model will be used to analyze development of new severe symptoms.
Early Treatment Upamostat Arm: Proportion of participants who report: - Return to usual state of health - Return to usual activities | Days 7, 14, 28, Week 8, and Week 12
  A Cox proportional hazards model will be used to analyze the time to: - return to usual state of health - return to usual activities.
Early Treatment Upamostat Arm: Proportion of participants hospitalized for COVID-19 | Day 0 to Week 12
  Adjudicated prior to study unblinding.
Early Treatment Upamostat Arm: Number and proportion of participants hospitalized (all cause) | Day 0 to Day 28
Early Treatment Upamostat Arm: Number and proportion of participant deaths (all cause) | Day 0 to Day 28
Early Treatment Upamostat Arm: Comparison of active and placebo treatment groups in time to negative PCR | Day 0 to Week 12
  Time to negative RT-PCR will be defined as the time of the first of two consecutive readings below the lower limit of detection. A Cox proportional hazards model will be used to analyze the time to negative PCR.

OTHER OUTCOMES:
Early Treatment Upamostat Arm: Incidence of Serious Adverse Events (SAE) | Day 0 to Week 12
Early Treatment Upamostat Arm: Comparison between active and placebo treatment groups in proportion of all and greater than or equal to grade 3 adverse events. | Day 0 to Week 12
  Assessed by the National Institutes of Health, Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table), corrected Version 2.1, July 2017
Early Treatment Upamostat Arm: Incidence of AEs causing IP discontinuation | Day 0 to Week 12
Early Treatment Upamostat Arm: Incidence of all-cause IP discontinuation or interruption | Day 0 to Week 12
Early Treatment Upamostat Arm: Number of participants hospitalized due to adverse events regardless of cause | Day 0 to Week 12
Early Treatment Upamostat Arm: Difference in proportion of participants meeting the primary endpoint between treatment and placebo by variant of concern (VOC) via viral genome sequencing. | Day 0 to Week 12
Early Treatment Upamostat Arm: Number and proportion of participants with anti-SAR-CoV2 IgM antibodies by treatment assignment | Day 0 and Week 8
  Difference in anti-SARS-CoV2 IgM geometric mean antibody titers among antibody positive patients by treatment assignment
Early Treatment Upamostat Arm: Number and proportion of participants with anti-SAR-CoV2 IgG antibodies by treatment assignment | Day 0 and Week 8
  Difference in anti-SARS-CoV2 IgG geometric mean antibody titers among antibody positive patients by treatment assignment
Early Treatment Upamostat Arm: Number and proportion of patients with certain targeted polymorphisms in host transmembrane proteases by treatment group and outcome. | Day 0 to Week 12

CONTACTS AND LOCATIONS:
Locations (6):
- United States (3):
  - Johns Hopkins Hospital, Baltimore, Maryland
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - KUR Research, Nashville, Tennessee
- Josha Research, Bloemfontein, South Africa
- Royal Thai Army Clinical Research Center (RTA CRC) Royal Thai Army-Armed Forces Research Institute of Medical Sciences (RTA-AFRIMS), Bangkok, Thailand
- Makerere University Walter Reed Project, Fort Portal, Uganda

IPD SHARING:
Plan to Share IPD: Undecided